CLINICAL TRIAL: NCT02305368
Title: Evaluation of Interest Chemo-oncogramme in Patients With Colonic Adenocarcinoma Stage 4: a Pilot Study
Brief Title: Evaluation of Interest Chemo-oncogramme in Patients With Colonic Adenocarcinoma Stage 4
Acronym: Oncogramme
Status: Completed | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: I09019 Oncogramme colon
Record Dates: First submitted 2014-11-19; First posted 2014-12-02 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — tumor fragment
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Oncogramme: Taking a fragment of colon tumors taken from a specimen. Cells fragment are cultured for 7 days. The effects of chemotherapy are studied on these cells through chimio-oncogramme.
  Interventions: Other: Chimio-oncogramme

INTERVENTIONS:
Other: Chimio-oncogramme — Cells fragment are cultured for 7 days. The effects of chemotherapy are studied on these cells through chimio-oncogramme.

SUMMARY:
In patients with colonic adenocarcinoma stage 4 which are potentially resectable metastases (lung and liver metastases), treatment with chemotherapy is necessary but not end in success in 10% of cases. The development of techniques for administering personalized treatment becomes necessary for these patients. Thus, in vitro tests on cells from tumors of these patients and evaluating the effect of chemotherapy on these could be made for each patient. In France, the company develops Oncomedics these tests.

This is a pilot study that will make a first evaluation under actual conditions of chimio-oncogramme.

DETAILED DESCRIPTION:
A fragment of colon tumors will be taken from a specimen or a cold biopsy, tissue from patients diagnosed with colon carcinoma metastatic (stage 4). In parallel and systematically: analysis by the pathologist of a histological section.

* Culturing the cells obtained from the tumor by Oncomedics fragment in a defined medium and provided for enriching tumor cells compared to stromal cells.
* Maintaining the cells in culture for 7 days.
* Effects of conventional chemotherapy (corresponding to protocols) on these cells for 72 hours (growth chambers) by Oncomedics (chimio-oncogramme).
* For each chemotherapy tested, measuring the proportion of dead cells / total cells.
* Retained by Oncomedics results, not given to the nursing team. The patient will be treated and followed up in the usual way.
* At the end of the study, comparing the in vitro results (chimio-oncogramme) to the patient's response to (x) the same (s) chemotherapy (s).

ELIGIBILITY:
Inclusion Criteria:

* patient with adenocarcinoma of the colon diagnosed at stage 4 receiving standard therapy
* targets must be measurable tumor lesions (RECIST)
* patient has not expressed opposition to the use of their residual tumor

Exclusion Criteria:

* Against-formal indication to an indispensable para-clinical examination of the patient monitoring
* Use of chemotherapy, hormone therapy or concomitant radiotherapy
* Cons-indication for chemotherapy
* Are pregnant, nursing or lack of contraception for women of childbearing age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient with adenocarcinoma of the colon diagnosed at stage 4 receiving standard therapy
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2011-03; Primary Completion 2012-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
In vitro analysis of chemotherapy responses | 7 days
  Evaluate the predictive value of chemo-oncogramme on the patient's response to the same (s) chemotherapy (s)

SECONDARY OUTCOMES:
quality of life | 7 days
  Evaluate the predictive value of chemo-oncogramme on chemical toxicity and quality of life of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Muriel MATHONNET, MD, Principal Investigator — Chirurgie digestive - CHU LIMOGES

REFERENCES:
- [Derived] Bounaix Morand du Puch C, Nouaille M, Giraud S, Labrunie A, Luce S, Preux PM, Labrousse F, Gainant A, Tubiana-Mathieu N, Le Brun-Ly V, Valleix D, Guillaudeau A, Mesturoux L, Coulibaly B, Lautrette C, Mathonnet M. Chemotherapy outcome predictive effectiveness by the Oncogramme: pilot trial on stage-IV colorectal cancer. J Transl Med. 2016 Jan 12;14:10. doi: 10.1186/s12967-016-0765-4. PMID 26791256